CLINICAL TRIAL: NCT05582642
Title: Respiratory Muscles After Inspiratory Muscle Training in Patients After COVID-19 With Persistent Dyspnea and Respiratory Muscle Dysfunction
Brief Title: Respiratory Muscles After Inspiratory Muscle Training After COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Jens Spießhöfer, Principal Investigator, RWTH Aachen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTCA 250-22 / 22-241
Record Dates: First submitted 2022-10-09; First posted 2022-10-17 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: COVID-19; Diaphragm Injury
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diaphragm Strength Training (Active Comparator)
  Interventions: Device: Inspiratory Muscle Training (IMT)
- Diaphragm Endurance Training (Sham Comparator)
  Interventions: Device: Inspiratory Muscle Training (IMT)

INTERVENTIONS:
Device: Inspiratory Muscle Training (IMT) — The training itself includes 2 x 30 breathing cycles per day. The whole training should take place daily, 7 days a week. The initial training intensity in the treatment arm (resistance of the respiratory muscle training) is set to 50% of the maximum respiratory muscle strength (measured using PImax). Once a week the present investigators get a picture of patient's training, pay attention to shortness of breath, potential for adaptation.
  In the "control" arm of the study, this force adjustment would not take place, i.e. it is an endurance training of the diaphragm (10% of PI Max over the whole 6 weeks) with, however, also the control dates of the training twice a week. At least in the 6 weeks of the study (see above).

SUMMARY:
It is the aim of the current (follow-up) project for the first time in post-COVID-19 patients who continue to complain of shortness of breath and for whom there is no other explanation than possibly proven diaphragmatic weakness, to determine the effects of 6 weeks of IMT/diaphragm training on diaphragm strength and shortness of breath.

DETAILED DESCRIPTION:
Breathing is a complex process involving muscular, neurological and chemical processes in the body. Herein, the respiratory muscles play a very important role.

The respiratory muscles are the muscle groups that cause the expansion and contraction of the chest during inhalation and exhalation. The most important respiratory muscle is the diaphragm. It is known that long-term ventilation in the intensive care unit weakens the respiratory muscles, since the work of the muscles is taken over by the ventilation devices and the muscles are not trained over a long period of time.

As recently shown, COVID-19 disease can lead to diaphragmatic weakness even in the absence of ventilation.

In this project (CTCA 20-515) the present investigators demonstrated that several patients after COVID-19 suffer from diaphragmatic weakness. Specifically, diaphragmatic weakness also related to shortness of breath complained about by patients and currently not otherwise explainable.

The so-called inspiratory muscle training (IMT or diaphragm training) is known in pneumological rehabilitation for years. In the current project, after the training has been explained, the patient is asked to breathe against resistance at home using a small mouthpiece and a small device several times (twice) a day and several times a week (each day).

This procedure is considered safe and very effective in training the diaphragm. Accordingly, it is the aim of the current (follow-up) project for the first time in post-COVID patients who continue to complain of shortness of breath and for whom there is no other explanation than possibly the proven diaphragmatic weakness, to determine the effects of 6 weeks of IMT/diaphragm training on diaphragm strength and on shortness of breath.

At the beginning and at the end of the 6 weeks of training, the present investigators would carry out the all-encompassing measurement of diaphragm force, which is known to patients and explained again below. Furthermore, the present investigators would invite patients twice a week to optimize the training together (for a maximum of 1 hour per appointment). This would take place once a week in the present investigators laboratory for respiratory physiology and the training would be improved it if necessary, once a week.

The training would end after 6 weeks and the present investigators would measure diaphragm function again 6 weeks after the training, i.e. a third time in total, to determine whether the effects seen continue to be present after the training. After that, the study ends.

The present investigators would offer the treatment arm (the 9/18 patients) in whom diaphragm endurance training was carried out as a control of the diaphragmatic strength training to carry out strength training after the measurement 6 weeks after the end of the therapy (outside of this study here as a purely clinical therapy).

The training itself includes 2 x 30 breathing cycles per day. Patients can divide these 2 x 30 breathing cycles freely, i.e. specifically train 1 x 30 breathing cycles in the morning and 1 x 30 breathing cycles in the afternoon. The whole training should take place daily, 7 days a week.

Once a week the present investigators get a picture of the patient's training, pay attention to shortness of breath, potential for adaptation (also specifically for even stronger training, if tolerated by the patients, increase in training, i.e. the breathing resistance that patients would have to overcome when inhaling ).

In the "control" arm of the study, this force adjustment would not take place, i.e. it is an endurance training of the diaphragm with, however, also the control dates of the training twice a week. At least in the 6 weeks of the study (see above).

ELIGIBILITY:
Inclusion Criteria:

* 18 patients with survived COVID-19, persistent otherwise unexplainable dyspnoea and proven diaphragm dysfunction
* Patients aged at least 18 years, who are mentally and physically able to consent and participate into the study

Exclusion Criteria:

* Diagnosis of another disease, which causes a permanent increase in carbon dioxide level in the blood (chronic hypercapnia) or a permanent combined lung weakness (particularly a neuromuscular disease)
* Body-mass-index (BMI) >40
* Expected absence of active participation of the patient in study-related measurements
* Alcohol or drug abuse
* Metal implant in the body that is not MRI compatible (NON MRI compatible pacemaker, implantable defibrillator, cervical implants, e.g. brain pacemakers etc.)
* Slipped disc
* Epilepsy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Twitch transdiaphragmatic pressure in response to supramaximal magnetic stimulation of the phrenic nerve roots (Unit: Pressure in cmH2O) | Assessed at baseline
Twitch transdiaphragmatic pressure in response to supramaximal magnetic stimulation of the phrenic nerve roots (Unit: Pressure in cmH2O) | Assessed after 6 weeks of IMT
Twitch transdiaphragmatic pressure in response to supramaximal magnetic stimulation of the phrenic nerve roots (Unit: Pressure in cmH2O) | Assessed 6 weeks after IMT
Respiratory mouth pressures | Assessed at baseline
  Measurement of respiratory (inspiratory and expiratory) mouth pressures (Unit: Pressure in cmH2O)
Respiratory mouth pressures | Assessed after 6 weeks of IMT
  Measurement of respiratory (inspiratory and expiratory) mouth pressures (Unit: Pressure in cmH2O)
Respiratory mouth pressures | Assessed 6 weeks after IMT
  Measurement of respiratory (inspiratory and expiratory) mouth pressures (Unit: Pressure in cmH2O)

SECONDARY OUTCOMES:
Diaphragm and Intercostal ultrasound | Assessed at baseline
  Thickening fraction (Unit: %)
Diaphragm and Intercostal ultrasound | Assessed after 6 weeks of IMT
  Thickening fraction (Unit: %)
Diaphragm and Intercostal ultrasound | Assessed 6 weeks after IMT
  Thickening fraction (Unit: %)
Exercise intolerance | Assessed at baseline
  Dyspnea (Borg dyspnea scale; Unit 1-10 with higher values indicating more severe dyspnea)
Exercise intolerance | Assessed after 6 weeks of IMT
  Dyspnea (Borg dyspnea scale; Unit 1-10 with higher values indicating more severe dyspnea)
Exercise intolerance | Assessed 6 weeks after IMT
  Dyspnea (Borg dyspnea scale; Unit 1-10 with higher values indicating more severe dyspnea)
Lung function | Assessed at baseline
  Comprehensive assessment of lung function (most importantly forced vital capacity; Unit Liters)
Lung function | Assessed after 6 weeks of IMT
  Comprehensive assessment of lung function (most importantly forced vital capacity; Unit Liters)
Lung function | Assessed 6 weeks after IMT
  Comprehensive assessment of lung function (most importantly forced vital capacity; Unit Liters)
Electromyography of diaphragm and accessory respiratory muscle activity | Assessed at baseline
  Activity of the respiratory muscles (Unit: % with higher values indicating higher activity of the respiratory muscles)
Electromyography of diaphragm and accessory respiratory muscle activity | Assessed after 6 weeks of IMT
  Activity of the respiratory muscles (Unit: % with higher values indicating higher activity of the respiratory muscles)
Electromyography of diaphragm and accessory respiratory muscle activity | Assessed 6 weeks after IMT
  Activity of the respiratory muscles (Unit: % with higher values indicating higher activity of the respiratory muscles)

CONTACTS AND LOCATIONS:
Overall Officials: Jens Spiesshoefer, MD, Principal Investigator — RWTH Aachen University; Binaya Regmi, MD, Study Chair — RWTH Aachen University; Michael Dreher, Professor, Study Director — RWTH Aachen University
Locations (1):
- RWTH Aachen University, Aachen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Daher A, Balfanz P, Aetou M, Hartmann B, Muller-Wieland D, Muller T, Marx N, Dreher M, Cornelissen CG. Clinical course of COVID-19 patients needing supplemental oxygen outside the intensive care unit. Sci Rep. 2021 Jan 26;11(1):2256. doi: 10.1038/s41598-021-81444-9. PMID 33500431
- [Background] Daher A, Balfanz P, Cornelissen C, Muller A, Bergs I, Marx N, Muller-Wieland D, Hartmann B, Dreher M, Muller T. Follow up of patients with severe coronavirus disease 2019 (COVID-19): Pulmonary and extrapulmonary disease sequelae. Respir Med. 2020 Nov-Dec;174:106197. doi: 10.1016/j.rmed.2020.106197. Epub 2020 Oct 20. PMID 33120193
- [Background] Balfanz P, Hartmann B, Muller-Wieland D, Kleines M, Hackl D, Kossack N, Kersten A, Cornelissen C, Muller T, Daher A, Stohr R, Bickenbach J, Marx G, Marx N, Dreher M. Early risk markers for severe clinical course and fatal outcome in German patients with COVID-19. PLoS One. 2021 Jan 29;16(1):e0246182. doi: 10.1371/journal.pone.0246182. eCollection 2021. PMID 33513168
- [Background] Spiesshoefer J, Friedrich J, Regmi B, Geppert J, Jorn B, Kersten A, Giannoni A, Boentert M, Marx G, Marx N, Daher A, Dreher M. Diaphragm dysfunction as a potential determinant of dyspnea on exertion in patients 1 year after COVID-19-related ARDS. Respir Res. 2022 Jul 15;23(1):187. doi: 10.1186/s12931-022-02100-y. PMID 35841032
- [Result] Spiesshoefer J, Henke C, Herkenrath S, Brix T, Randerath W, Young P, Boentert M. Transdiapragmatic pressure and contractile properties of the diaphragm following magnetic stimulation. Respir Physiol Neurobiol. 2019 Aug;266:47-53. doi: 10.1016/j.resp.2019.04.011. Epub 2019 Apr 25. PMID 31029769
- [Result] Spiesshoefer J, Henke C, Herkenrath S, Randerath W, Brix T, Young P, Boentert M. Assessment of Central Drive to the Diaphragm by Twitch Interpolation: Normal Values, Theoretical Considerations, and Future Directions. Respiration. 2019;98(4):283-293. doi: 10.1159/000500726. Epub 2019 Jul 26. PMID 31352459
- [Result] Spiesshoefer J, Herkenrath S, Henke C, Langenbruch L, Schneppe M, Randerath W, Young P, Brix T, Boentert M. Evaluation of Respiratory Muscle Strength and Diaphragm Ultrasound: Normative Values, Theoretical Considerations, and Practical Recommendations. Respiration. 2020;99(5):369-381. doi: 10.1159/000506016. Epub 2020 May 12. PMID 32396905
- [Derived] Spiesshoefer J, Regmi B, Senol M, Jorn B, Gorol O, Elfeturi M, Walterspacher S, Giannoni A, Kahles F, Gloeckl R, Dreher M. Potential Diaphragm Muscle Weakness-related Dyspnea Persists 2 Years after COVID-19 and Could Be Improved by Inspiratory Muscle Training: Results of an Observational and an Interventional Clinical Trial. Am J Respir Crit Care Med. 2024 Sep 1;210(5):618-628. doi: 10.1164/rccm.202309-1572OC. PMID 38763165